CLINICAL TRIAL: NCT00266786
Title: A Phase 3, Double-Blind, Randomized Study of the Safety, Tolerability, and Analgesic Efficacy of Multiple Doses of Ketorolac Tromethamine Administered Intranasally for Postoperative Pain Following Major Abdominal Surgery
Brief Title: Safety and Efficacy of Multiple Doses of Intranasal Ketorolac in Postoperative Pain Following Major Abdominal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: David Bregman, M.D., Ph.D., Luitpold Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROX 2005-01
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Intranasal Ketorolac Tromethamine (Experimental)
  Interventions: Drug: Intranasal Ketorolac Tromethamine
- Intranasal Placebo (Placebo Comparator)
  Interventions: Drug: Intranasal Placebo

INTERVENTIONS:
Drug: Intranasal Ketorolac Tromethamine — Intranasal at 30mg
  Arms: Intranasal Ketorolac Tromethamine
Drug: Intranasal Placebo — Intranasal Placebo
  Arms: Intranasal Placebo

SUMMARY:
Ketorolac has been marketed for several years in other forms (tablet and injectable) for the short-term relief of pain. This study will test whether a new dosage form (nasal spray) containing ketorolac is effective at relieving the pain of major abdominal surgery, and will also assess product safety. Previous studies with the nasal spray have suggested that it is similar to the previously approved injectable form in effectiveness for pain relief and in its safety profile.

Patients will be randomized in a 2:1 ratio to receive intranasal ketorolac or placebo when the pain reaches a moderate level (40 on a scale of 100) following surgery. After the first dose, subjects will receive study drug every 6 hours for 48 hours, and then as needed (up to 4 times a day) for a total of 5 days. If pain is not adequately relieved by the study drug, subjects will be given morphine sulfate or other standard analgesics. Follow-up safety evaluations will occur about 1 and 2 weeks after the start of dosing.

Subjects will be asked to answer questions about their pain relief and any possible side effects of the drug during the study, and will be given physical examinations, including nasal evaluations, before and during the clinical trial. A small amount of blood will be drawn for routine clinical laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18 through 64 years
* Major abdominal surgery
* Body weight ≥ 100 and ≤ 300 pounds
* Negative serum pregnancy test
* Pain intensity score at least 40 (moderate pain) on 100 mm visual analog scale
* Minimum 48 hour hospital stay and 5 day maximum stay
* Able to provide written informed consent
* Willing and able to comply with all testing requirements of the protocol

Exclusion Criteria:

* Allergy or sensitivity to ketorolac or ethylene diamine tetraacetic acid (EDTA)
* Allergy or significant reaction to opioids
* Allergic reaction to aspirin or other nonsteroidal anti-inflammatory drug (NSAIDs)
* Current upper respiratory tract infection or other respiratory tract condition that could interfere with absorption of the nasal spray or adverse event assessment
* Use of any intranasal product in past 24 hours
* Clinically significant abnormality on screening lab tests
* History of cocaine use
* Active peptic ulcer disease or significant history of peptic ulcer disease or gastrointestinal bleeding
* Advanced renal impairment or risk for renal failure
* History of other medical problems that could interfere with the study participation
* Pregnancy or breastfeeding
* Participation in another investigational study within past 30 days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 321 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The Summed Pain Intensity Difference (SPID) on Day 1 | 6 hours after drug administration
  Ratings of Pain Intensity (PI) were made using a 100-mm Visual Analog Scale (VAS) on which 0 = no pain and 100 = worst pain possible. The PI values were obtained every hour following the first dose of study medication on Day 1. Pain intensity difference (PID) was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication. A summed PID (SPID) on the first postoperative day was calculated at 6 hours.

SECONDARY OUTCOMES:
Pain intensity difference scores | Prior to receiving study drug and at 20, 40, and 60 minutes, and 2, 3, 4, 5, 6, 12, 18, 24, 30, 36, 42, and 48 hours after the first dose, then prior to each dose up to 72 hours
  Ratings of Pain Intensity (PI) were made using a 100-mm Visual Analog Scale (VAS) on which 0 = no pain and 100 = worst pain possible. PID was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication.
Quality of analgesia | Prior to receiving study drug and at 20, 40, and 60 minutes, and 2, 3, 4, 5, 6, 12, 18, 24, 30, 36, 42, and 48 hours after the first dose, then prior to each dose up to 72 hours
  Quality of analgesia was assessed on a 5-point categorical scale with 0 = poor, 1 = fair, 2 = good, 3 = very good, and 4 = excellent.
Global assessment of pain control | 8 hours following first dose of study medication
  A global evaluation of pain control was conducted once daily at bedtime using a 5-point categorical scale on which 0 = poor, 1 = fair, 2 = good, 3 = very good, and 4 = excellent.
Morphine sulfate consumption at 24, 48, and 72 hours | 24, 48, and 72 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln Bynum, MD, Study Chair — ICON Clinical Research
Locations (6):
- United States (5):
  - Methodist Hospital, Arcadia, California
  - Glendale Adventist Medical Center, Glendale, California
  - Clinical Management Services, Inc., Pasadena, California
  - Memorial Hermann Healthcare System, Houston, Texas
  - Houston Perinatal Associates, Houston, Texas
- Waikato Clinical Research, Hamilton, New Zealand